CLINICAL TRIAL: NCT04076527
Title: Prospective, Multicenter Cohort Study on Primary Biliary Cholangitis
Acronym: PBC-Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Collaborators: RWTH Aachen University (Other); Zentrum für Klinische Studien Leipzig (Other); Intercept Pharma Europe Limited (IPEL) (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Hospital Erlangen (Other); Medical care center for Gastroenterology, Berlin (Unknown); Institute for Interdisciplinary Medicine, Hamburg (Unknown); Leberhilfe Projekt gUG, Cologne (Unknown); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Thomas Berg, Prof. Dr. Thomas Berg, University of Leipzig
Other Study IDs: 2.0
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: PBC; Primary Biliary Cholangitis
Keywords: ursodeoxycholic acid; UDCA; obeticholic acid; OCALIVA; Cohort; observational study; Bezafibrat; Budesonide
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid; obeticholic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 - Incomplete Responder: 1. Primary Incomplete Responder: PBC patients demonstrating an insufficient response to the standard therapy with ursodeoxycholic acid (UDCA) after a minimum of 12 months of treatment (Paris II criteria).
  2. Secondary Incomplete Responder: PBC patients demonstrating a satisfactory initial response to UDCA after a minimum of 12 months of treatment (Paris II criteria) followed by a re-increase of ALP ≥1.5 ULN, or AST ≥1.5 ULN, or bilirubin >1 mg/dl at any later time point during continuous UDCA-treatment.
  Interventions: Drug: UDCA; Drug: Ocaliva
- Group 2 - Responder: PBC patients demonstrating a satisfactory initial and contin-ued response to UDCA after a minimum of 12 months of treatment (Paris II criteria) without a re-increase of ALP ≥1.5 ULN, or AST ≥1.5 ULN, or bilirubin >1 mg/dl at any later time point during continuous UDCA-treatment.
  Interventions: Drug: UDCA
- Group 3: Patients newly diagnosed for PBC receiving an approved PBC therapy for the first time. Patients are considered to be newly diagnosed if the initial diagnosis took place no later than six months prior to inclusion into the study.
  Interventions: Drug: UDCA; Drug: Ocaliva

INTERVENTIONS:
Drug: UDCA — Routine data is collected for UDCA therapy.
  Other Names: ursodeoxycholic acid
Drug: Ocaliva — Routine data is collected for OCA therapy.
  Other Names: obeticholic acid
  Groups: Group 1 - Incomplete Responder; Group 3

SUMMARY:
The German PBC Cohort is a multi-centric, observational (non-interventional) study with three parallel groups. The main objective of this observational study is to describe the course of Primary biliary cholangitis (PBC) in patients in Germany under routine treatment with approved drugs. Therefore, the effectiveness and safety/tolerability of PBC treatment options in a real-life setting will be evaluated.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC) is a chronic autoimmune cholestatic liver disease. The course of the disease is characterized by a slow destruction of bile ducts, and progressive cholestasis. Prognosis depends on the development of cirrhosis and its complications. Ursodeoxycholic acid (UDCA) has been established as standard therapy for PBC and improves patients' long-term outcome. However, UDCA is not a uniformly effective drug, and the prognosis of PBC patients insufficiently responding to treatment is markedly worse. For patients with suboptimal treatment response to UDCA obeticholic acid (OCA) as newly approved medication (OCALIVA®) is available as second line treatment.

Due to the low prevalence and the slowly progressive course of the disease it is very difficult to investigate the prognosis of subgroups of PBC patients or to evaluate the effectivness of therapeutic interventions on clinical outcomes. Therefore, several national or international registries (UK-PBC Consortium or the Global PBC Study Group) were founded to better characterize the clinical course of PBC patients.

Since in Germany a registry for PBC does not exist, the German PBC Cohort is being implemented as observational study to collect data on treatment progress and success in clinical routine that reflects real world conditions in Germany as closely as possible. The effectiveness and safety/tolerability of PBC treatment options (UDCA as standard therapy and second-line treatment options like OCALIVA in case of inadequate UDCA treatment response) will be evaluated.

In approximatly 40 sites in Germany routine data is collected. There are no specifications for the diagnosis, therapy and monitoring of the PBC patients. The documentation of the routine data is carried out alongside with guideline recommended treatment intervals of the patients.

Furthermore, a critical criterion for the German PBC Cohort study is the involvement of a sufficient number of gastroenterology specialized practices and outpatient clinics that have consciously not been selected based on the strict specifications of a clinical trial and which provide routine treatment for PBC patients. In addition, patient access is designed to be open. Data will be collected on patient groups that represent a majority of the PBC patients in Germany, but who are not being investigated in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of PBC PBC diagnosis (consistent with AASLD and EASL practice guidelines), as demonstrated by the presence of at least two of the following three diagnostic factors:

   * History of elevated ALP levels for 6 months.
   * Positive anti-mitochondrial antibody (AMA) titer or if AMA negative or in low titer (<1:80) => PBC-specific antibodies:

     * anti-GP210 and/or
     * anti-SP100 and/or
     * antibodies against the major M2 components [PDC-E2, 2-oxo-glutaric acid dehydrogenase complex (OADC-E2), branched-chain-2-oxo-acid-dehydrogenase complex, (BCOADC-E2)].
   * Liver biopsy consistent with PBC.
3. Medication-based treatment with at least one drug approved in Germany for the treatment of PBC
4. Availability of all following essential parameters at the initial diagnosis of PBC prior to the initiation of treatment with UDCA, 12 months after initiation of UDCA and if applicable at time point of secondary incomplete response:

   * Platelet count
   * Alkaline Phosphatase (ALP)
   * Total Bilirubin
   * Aspartate aminotransferase (AST/GOT)
   * Age at initial diagnosis of PBC
5. Patients must meet criteria of one of the cohorts (group 1/2/3) within this NIS according to design
6. written statement of informed consent

Exclusion Criteria:

Current participation in a phase I to IV interventional clinical trial for PBC or participation in another PBC registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited in gastroenterology specialized practices and outpatient clinics which provide routine treatment for PBC patients.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Systematic registry | from baseline to 36 months after baseline (observational period)
  A primary outcome measure is not applicable as usual, since this data acquisition is performed to built a newly developed systematic registry which serves to describe - for the first time in Germany - the characteristics and the recent state of usual clinical care of the respective population.
  Within the 18 months of recruitment and 3 years of individual follow-up for every patient regular analyses will be performed and published, based on a statistical analysis plan which may be yearly updated on request to address the main questions of the responsible PBC consortium.
  After the end of data acquisition hepatologic scientists may apply with detailed proposals to further use available data. A scientific consortium will than decided on further analyses of data.

SECONDARY OUTCOMES:
Comprehensive clinical characterization of German PBC patients | from baseline to 36 months after baseline
  i.e. demographics, biochemical markers, ultrasound, transient elastography, stage of the disease
Characterization of PBC therapies | from baseline to 36 months after baseline
  Characterization of UDCA as first line therapy and characterization of approved second-line treatment options such as OCALIVA.
  Furthermore, safety data on the PBC medications used will be systematically gathered and reported on high-level aggregation with regard to any causality with PBC treatment per cohort. The respective results will be reviewed against the known safety profiles.
Treatment response to PBC therapies after 12 months and during longer courses of application | from baseline to 12 months after baseline and to 36 months after baseline
  To evaluate the natural progression under PBC drug therapy with respect to response to treatment changes in laboratory results (as ratios of the upper/lower limits of normal or differences to BL values) and characteristics of liver function will be described, e.g.:
  1. frequency of hepatic decompensation (occurrence of variceal hemorrhage, ascites, encephalopathy, and/or hepatocellular carcinoma),
  2. frequency of liver transplants,
  3. frequency of deaths in total and from a liver-related cause, and
  4. details on further events of special interest, e.g. for the first time serum bilirubin > ULN and/or alkaline phosphatase > 1.5 ULN, or transient elastography > 9.6 kPa.
Application and analyses of existing prognostic PBC scores to provide information on patients' prognosis. | from baseline to 36 months after baseline
  Details on typical therapeutic measures in treating PBC and patient compliance will be presented. This allows making a statement on quality of PBC treatment in Germany. Effectiveness will be assessed per cohort and compared between physicians' practices and hospital outpatient departments, aggregating data over all participating sites of the respective structure of health care. This refers to GLOBE score and/or Paris II criteria, frequency of hepatic decompensation or frequency of abnormal surrogate parameter (i.e. alkaline phosphatase, bilirubin, ALAT, ASAT or transient elastography). The respective results will be discussed against the results provided from clinical trials to verify everyday suitability of the different PBC therapies.
Concomitant Medications | from baseline to 36 months after baseline
  Assessment of selected concomitant medications (e.g. symptomatic treatment of pru-ritus)
Concomitant Autoimmune Diseases | from baseline to 36 months after baseline
  Assessment of selected concomitant autoimmune diseases (e.g. overlap syndrome with autoimmune hepatitis)
Concomitant Non-Autoimmune Diseases | from baseline to 36 months after baseline
  Assessment of selected concomitant non-autoimmune diseases (i.e. cardiovascular disease, non-alcoholic fatty liver disease, metabolic syndrome, chronic kidney diseases)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berg, Prof.Dr., Study Chair — University of Leipzig; Johannes Wiegand, Prof.Dr., Principal Investigator — University of Leipzig; Christian Trautwein, Prof.Dr., Principal Investigator — RWTH Aachen University
Locations (50):
- Germany (50):
  - University Hospital Aachen, Aachen
  - Charité - Campus Benjamin Franklin, Berlin
  - Charité-Campus Virchow-Klinikum, Berlin
  - Internal Practice, Berlin
  - Liver Center Checkpoint, Berlin
  - MVZ Gastroenterology, Berlin
  - Hospital Chemnitz, Chemnitz
  - University Hospital Cologne, Cologne
  - Internal Practice, Dornstadt
  - MVZ Düsseldorf, Düsseldorf
  - University hospital Düsseldorf, Düsseldorf
  - University Hospital Erlangen, Erlangen
  - St. Josef- Hospital Kupferdreh, Essen
  - University Hospital Essen, Essen
  - Internal Practice, Frankfurt
  - University Hospital J.W. Goethe- Universität, Frankfurt am Main
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Gießen, Giessen
  - Gastroenerological-Oncological Practice, Halle
  - University Hospital Halle, Halle
  - Liver Center Hamburg - Asklepios Clinic St. Georg, Hamburg
  - Internal Practice, Hamelin
  - MHH, Hanover
  - University Hospital Heidelberg, Heidelberg
  - Gastroenerological Practice, Herne
  - University hospital Saarland, Homburg
  - University Hospital Jena, Jena
  - Gastroenerological Practice, Kassel
  - Center for Gastroenterology and Hepatology Kiel, Kiel
  - University Hospital Schleswig-Holstein Campus Kiel, Kiel
  - Eugastro - Gastroenerological Practice, Leipzig
  - University Hospital Leipzig, Leipzig
  - MVZ Leverkusen, Leverkusen
  - University hospital Schleswig-Holstein, Lübeck
  - Internal Practice Hepatology, Magdeburg
  - University hospital Magdeburg, Magdeburg
  - University Hospital Mainz, Mainz
  - University Hospital Mannheim, Mannheim
  - Hospital LMU, Munich
  - Liver Center Munich, Munich
  - Technical University - Klinikum rechts der Isar, Munich
  - University Hospital Münster, Münster
  - Hospital Nuremberg, Nuremberg
  - Internal Practice, Potsdam
  - University Hospital Regensburg, Regensburg
  - Diakonie-Klinikum Schwäbisch Hall, Schwäbisch Hall
  - Internal Practice, Schwerin
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - St. Josefs-Hospital, Wiesbaden

IPD SHARING:
Plan to Share IPD: Undecided